CLINICAL TRIAL: NCT02471638
Title: PQ Bypass Systems for Femoropopliteal Bypass II (PQB 4 FP II)
Brief Title: DETOUR I Clinical Study for Percutaneous Femoropopliteal Bypass
Acronym: DETOUR1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STP 115
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single arm study (Experimental): PQ Bypass System for Femoropopliteal Bypass to complete percutaneous fem-pop bypass
  Interventions: Device: PQ Bypass System for Femoropopliteal Bypass

INTERVENTIONS:
Device: PQ Bypass System for Femoropopliteal Bypass — To access, deliver guidewires and implant stent grafts for a percutaneous fem-pop bypass.

SUMMARY:
To assess the safety and performance of the PQ Bypass System to access, deliver guidewires and implant stent grafts for a percutaneous fem-pop bypass.

DETAILED DESCRIPTION:
Prospective, single-arm, multi-center, international, non-randomized, pre-market, safety and effectiveness clinical investigation evaluating the PQ Bypass Systems to access, deliver guidewires and implant stent grafts for a percutaneous femoropopliteal (fem-pop) bypass.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Age 18 or older
* Rutherford Classification of 3-5
* Patent iliac and femoral arteries/veins and access vessels, of sufficient size and morphology (including tortuosity), to allow endovascular access with 8 Fr. introducer sheath
* Femoro-popliteal lesions ≥10 cm in length considered to be:

  * Chronic total occlusion (100% stenosis)
  * Diffuse stenosis (>50% stenosis) with moderate to heavy calcification
  * In-stent restenosis (>50% stenosis)
* Proximal and distal target vessels are 5.4-7.0 mm in diameter
* Orifice and proximal 1 cm of SFA is patent
* Patent popliteal artery 3 cm proximal to tibial plateau
* At least 1 patent tibial artery to the foot
* Patent femoral vein ≥ 10 mm in diameter or duplicate femoral vein
* Subject has > one year life expectancy

Exclusion Criteria:

* Bypass length required > 30 cm
* History of deep vein thrombosis
* Has a known hypersensitivities, allergies or contraindications to: nitinol, PTFE; aspirin, heparin, antiplatelet, anticoagulant or thrombolytic therapy; or anticoagulation or contrast media that is not amenable to pre-treatment;
* Has a known history of intracranial bleeding or aneurysm, myocardial infarction or stroke within the last 12 months
* Pregnant or nursing
* Untreated flow-limiting aortoiliac occlusive disease
* Has renal failure (eGFR < 30mL/min)
* Major distal amputation (above the transmetatarsal) in the study or non-study limb
* Patient has had a revascularization procedure on the target limb within 30 days
* Patient has a planned amputation of the target limb
* Previous bypass surgery on the target limb
* Patient is participating in another clinical study for which follow-up is currently on going.
* Patient has a condition that in the view of the investigator precludes participation in this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, PhD, Principal Investigator — University of Leipzig
Locations (8):
- Universidad Católica de Chile, Santiago, Chile
- University of Leipzig Medical Centre, Leipzig, Germany
- Ospedale San Raffaele, Milan, Italy
- Stradins University Hospital, Riga, Latvia
- Vascular Service, Auckland, New Zealand
- Poland (3):
  - Gdansk Medical University, Gdansk
  - Poznan University of Medical Sciences, Poznan
  - Institute of Haematology Medicine Indira Gandhi, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schneider PA, Krievins DK, Halena G, Schmidt A, Lyden S, Lee V, Hu M, Adelman M. Venous outcomes at 1 year after using the femoral vein as a conduit for passage of percutaneous femoropopliteal bypass. J Vasc Surg Venous Lymphat Disord. 2021 Sep;9(5):1266-1272.e3. doi: 10.1016/j.jvsv.2020.12.080. Epub 2021 Jan 8. PMID 33429092
- [Derived] Krievins DK, Halena G, Scheinert D, Savlovskis J, Szopinski P, Kramer A, Ouriel K, Nair K, Holden A, Schmidt A. One-year results from the DETOUR I trial of the PQ Bypass DETOUR System for percutaneous femoropopliteal bypass. J Vasc Surg. 2020 Nov;72(5):1648-1658.e2. doi: 10.1016/j.jvs.2020.02.043. Epub 2020 Apr 8. PMID 32276015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 78 patients enrolled over the course of 24 months at 8 investigational sites
Units Other Than Participants: Lesions
Groups:
- Enrolled and Treated Patients: All patients enrolled in the DETOUR1 Clinical study to evaluate the PQ Bypass Detour System for Femoropopliteal Bypass to complete percutaneous fem-pop bypass.
  All patients were enrolled in the cath lab with a single procedure using the PQ Bypass Detour System, comprised of the PQ Crossing Device and the Torus Stent Graft System. Patients were followed to 24 months.
Period: Overall Study
Arm/Group | Enrolled and Treated Patients
Started | 78; 82 Lesions (One patient was enrolled but not treated due to technical failure of the device)
12 Month Results | 77; 79 Lesions
Completed | 68; 68 Lesions
Not Completed | 10; 14 Lesions
Not completed — Early Term Withdrawal | 10

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants enrolled 78, and Overall Number of Lesions (units) analyzed 82.
Units Other Than Participants: Lesions
Groups:
- Enrolled and Treated Patients: All patients and limbs enrolled in the DETOUR1 Study
Arm/Group | Enrolled and Treated Patients
Number analyzed (Participants) | 78
Number analyzed (Lesions) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 65
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: Lesions]
  New Zealand | 1
  Latvia | 34
  Poland | 36
  Italy | 1
  Chile | 7
  Germany | 3
Hypertension [Count of Participants; unit: Participants] | 65
Diabetes mellitus [Count of Participants; unit: Participants] | 20
Hypercholesterolemia [Count of Participants; unit: Participants] | 31
History of Coronary Artery Disease (CAD) [Count of Participants; unit: Participants] | 34
History of smoking [Count of Participants; unit: Participants] | 68
Previous peripheral vascular intervention [Count of Participants; unit: Participants] | 19
SFA lesion length [Mean (Standard Deviation); unit: mm] | 371 (55)
Ankle Brachial Index (ABI) [Mean (Standard Deviation); unit: Ratio] — Ankle Brachial Index is a measure of systolic blood pressure in the ankle divided by the systolic blood pressure in the brachial artery. lower ratios indicate a worse outcome. Ratios above 1.0 indicate non-compressible arteries
  Range measured at baseline in study- 0.34- 1.50
  Ratio | 0.64 (0.17)
TASC Lesion Type [Count of Units; unit: Lesions] — TASC II divides anatomic distribution of lesions into femoral popliteal. Lesion patterns are grouped into A-D lesions. TASC A lesions are those that should have excellent results from endovascular management. TASC B lesions are those that should have good results from endovascular management, and endoluminal interventions should be the first treatment approach. TASC C lesions are those for which surgical management provides superior long-term results and endovascular techniques should be reserved for patients who are surgically high risk. TASC D lesions should be treated by open surgery.
  Lesions
    TASC Lesion Type C | 46
    TASC Lesion Type D | 36
Chronic Total Occlusion [Count of Units; unit: Lesions] | 79
Rutherford Class [Count of Units; unit: Lesions] — Rutherford Classification is a system for grading clinical presentation of Peripheral Artery Disease (PAD)
  Classification 0- Asymptomatic-no hemodynamically significant occlusive disease Classification 1- Mild claudication Classification 2- Moderate claudication Classification 3- Severe claudication Classification 4- Ischemic rest pain Classification 5- Minor tissue loss-nonhealing ulcer, focal gangrene with diffuse pedal ischemia Classification 6- Major tissue loss-extending above Trans metatarsal level, functional foot no longer salvageable
  Lesions
    Rutherford Class 3 | 76
    Rutherford Class 4 | 5
    Rutherford Class 5 | 1
Calcification [Count of Units; unit: Lesions]
  Mild | 15
  Moderate | 11
  Severe | 55
  N/A | 1
Patent Tibial Runoff Vessels [Number; unit: Lesions] — The number of patent tibial arteries in the treated leg to carry blood flow to the lower leg and foot.
  Lesions
    1 | 6
    2 | 23
    3 | 49
    N/A | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions With Primary Patency
Description: Rate of primary patency. Primary patency defined as: no evidence of clinically significant stenosis (≥50%) within the stent graft or immediately above or below the treated arterial segment based on duplex ultrasound (systolic velocity ratio of >2.5).
Time Frame: 6 Months
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- Enrolled and Treated Patients: All limbs enrolled in the DETOUR1 Study
Arm/Group | Enrolled and Treated Patients
Number analyzed (Participants) | 78
Number analyzed (Lesions) | 81
Lesions | 72

2. Primary Outcome: Number of Lesions With Any Major Adverse Event (MAE) at One Month Post-procedure
Description: composite endpoint of death, CD-TVR, or major target limb amputation in all patients at One-month post procedure
Time Frame: One Month
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Groups:
- Enrolled Cohort: All limbs enrolled in the DETOUR1 Study
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 78
Number analyzed (Lesions) | 81
Lesions
  MAE | 2
  Free from MAE | 79

3. Secondary Outcome: Number of Lesions With Each Major Adverse Event (MAE) at One Month Post-procedure
Description: Outcome Measures of death, CD-TVR, or major target limb amputation as independent events one month post-procedure
Time Frame: One Month
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 78
Number analyzed (Lesions) | 81
Lesions
  Death | 0
  CD-TVR | 2
  Target Limb Amputation | 0
  Free from MAE | 79

4. Secondary Outcome: Percentage of Lesions With Primary Patency at 12 Months Post-Procedure
Description: Primary patency defined as: no evidence of clinically significant stenosis (≥50%) within the stent graft or immediately above or below the treated arterial segment based on duplex ultrasound (systolic velocity ratio of >2.5).
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 77
Number analyzed (Lesions) | 80
percentage of lesions | 81 (4)

5. Secondary Outcome: Major Adverse Vascular Event (MAVE) Rate
Description: Major Adverse Vascular Events-stent graft thrombosis, target limb amputation, clinically apparent distal embolization with tissue loss, procedure-related arterial rupture, acute limb ischemia, and bleeding events requiring any transfusion. Major bleeding required blood transfusion >2 units, and symptomatic deep vein thrombosis on ipsilateral limb
Time Frame: One Month
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 78
Number analyzed (Lesions) | 81
Lesions
  Stent thrombosis | 3
  Clinically apparent distal embolization | 0
  Procedure-related arterial rupture | 0
  Acute limb ischemia | 0
  Bleeding event requiring transfusion | 1
  Free from MAVE | 77
  Symptomatic Deep Vein Thrombosis on Ipsilateral Limb | 1

6. Secondary Outcome: Number of Lesions With Symptomatic Deep Vein Thromboses in Target Limb
Description: Rate of Symptomatic Deep Vein Thrombosis in target limb at one month time point.
Time Frame: One Month
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Enrolled and Treated Patients
Number analyzed (Participants) | 78
Number analyzed (Lesions) | 81
Lesions
  DVT in Target Limb | 1
  Freedom from DVT in Target Limb | 80

7. Secondary Outcome: Number of Major Adverse Events at the 12-Month Time Point
Description: Number of occurrences of all cause death, CD-TVR, or major target limb amputation
Time Frame: 12 Months
Measure: Number; unit: Events
Units Other Than Participants: Events
Groups:
- Enrolled Cohort: All limbs enrolled in the DETOUR1 Study that returned for 12M follow up
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 76
Number analyzed (Events) | 79
Events
  Death | 1
  CD-TVR | 12
  Target limb amputation | 0
  Freedom from MAE | 66

8. Secondary Outcome: Number of Major Adverse Events at the 3 Year Time Point
Description: Number of occurrences of all cause death, CD-TVR, or major target limb amputation
Time Frame: 3 Years
Measure: Number; unit: Events
Units Other Than Participants: Events
Groups:
- Enrolled Cohort: All patients that completed 3 year follow-up.
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 67
Number analyzed (Events) | 29
Events
  Death | 3
  Target limb amputation | 1
  CD-TVR | 27

9. Secondary Outcome: Major Adverse Vascular Event (MAVE) Rate at 3 Years
Description: as for outcome 5
Time Frame: 3 Years
Measure: Count of Participants; unit: Participants
Groups:
- Enrolled Cohort: All patients enrolled in the DETOUR1 Study
Arm/Group | Enrolled Cohort
Number analyzed (Participants) | 67
Participants
  Stent Graft Thrombosis (absence of TVR) | 15
  Clinically Apparent Distal Embolization | 0
  Procedure Related Arterial Rupture | 0
  Acute Limb Ischemia | 0
  Major Blood Loss Related to the PQ Bypass procedure requiring >2 units or packed RBC | 1
  Symptomatic Deep Vein Thrombosis on Ipsilateral Limb | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected at each follow-up visit through 3 years.
Groups:
- Enrolled and Treated Patients: All limbs enrolled in the DETOUR1 Study of the enrolled and treated patients.
  Some subjects had bilateral enrollment (the Detour Procedure was performed on both legs), because of this, the all-cause mortality rate has a different denominator than the other limb related adverse events. A total of 78 participants were enrolled (82 lesions), and one patient was enrolled but not treated due to technical failure of the device. The all-cause mortality denominators (at Risk values) are different from the other limb related adverse events. The all-cause mortality rate is reported at 1/77.
Arm/Group | Enrolled and Treated Patients
All-Cause Mortality (participants affected / at risk) | 3/78
Serious Adverse Events (participants affected / at risk) | 14/78
Other Adverse Events (participants affected / at risk) | 65/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled and Treated Patients (N=78)
Clinically Driven Target Vessel Revascularization (CD-TVR) (Surgical and medical procedures) | 12 (12) — Target Vessel Revascularization due to linically significant stenosis (≥50%) within the stent graft or immediately above or below the treated arterial segment based on duplex ultrasound (systolic velocity ratio of >2.5).
Target Limb Amputation (Surgical and medical procedures) | 0 (0)
Stent Thrombosis (Vascular disorders) | 13 (13)
Clinically apparent distal embolization (Vascular disorders) | 0 (0)
Procedure-related arterial rupture (Vascular disorders) | 0 (0)
Acute limb ischemia (Vascular disorders) | 0 (0)
Bleeding event requiring transfusion (Surgical and medical procedures) | 1 (1) — This event is subject specific, not lesion specific, therefore the number of participants at risk is adjusted
Deep Vein Thrombosis (DVT) (Vascular disorders) | 2 (2) — Deep Vein Thrombosis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enrolled and Treated Patients (N=78)
Access site hemorrhage or hematoma (Vascular disorders) | 3
Anemia (Blood and lymphatic system disorders) | 1
angina pectoris (Cardiac disorders) | 1
contralateral arteria femoral profunda occlusion (Vascular disorders) | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1
Bleeding Complications (Injury, poisoning and procedural complications) | 2 — Minor bleeding
Chronic Heart Failure (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Degenerative lumbar spondylosis (Musculoskeletal and connective tissue disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Deep Vein Thrombosis (Vascular disorders) | 4 — Not clinically significant
Drug Reaction (Injury, poisoning and procedural complications) | 3 — Mild Allergic reaction to contrast media or periprocedural medication
Edema (Blood and lymphatic system disorders) | 7 — Swelling
Stent Graft thrombosis (Vascular disorders) | 13
Fever (General disorders) | 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Diagnostic Hospitalization (Cardiac disorders) | 1
Stent Graft Occlusion (Vascular disorders) | 1
Arterio-Venous (A-V) Fistula between Posterior Tibial Artery (Injury, poisoning and procedural complications) | 1 — Other: A-V Fistula between Posterior Tibial Artery
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1
dislodgment of graft neo intima (General disorders) | 1
Endarteritis obliterans (Vascular disorders) | 1
Exacerbation of Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
Reflux (Vascular disorders) | 4
Hypertension (Vascular disorders) | 1
Hematoma (Injury, poisoning and procedural complications) | 1 — Patient received bruise on leg after fall in the garden
Occlusion of Contralateral Femoropopliteal Bypass (Vascular disorders) | 1 — Occlusion of Fem-pop bypass on contralateral limb
Stent Graft Migration (Injury, poisoning and procedural complications) | 1
Pain (General disorders) | 4 — Pain in Lower limbs
Stent Graft Stenosis (Vascular disorders) | 10
Rectal Bleeding (General disorders) | 1 — This Adverse event is calculated per patient, not per lesion, so the denominator reflects this difference
Reocclusion of bypass graft (Vascular disorders) | 1
Profundua Femoralis Stenosis (Vascular disorders) | 1 — Non target limb
Target Vessel Revascularization (TVR) (Vascular disorders) | 3
Arterial Ulcer (Vascular disorders) | 1 — Target Leg
transient ischemic attack (TIA) (Vascular disorders) | 1 — Transient Ischemic Attack

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT02471638/Prot_SAP_000.pdf